CLINICAL TRIAL: NCT04567290
Title: Pharmacodynamic Evaluation of Antiplatelet Effect of Swallowing Versus Chewing Ticagrelor in Patients With Acute Coronary Syndrome
Acronym: TICA-MASTICA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Hospitalario La Concepcion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2020-09-21; First posted 2020-09-28 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Ticagrelor; Platelet aggregation inhibitors; VerifyNow; Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chewed ticagrelor (Experimental): Ticagrelor pills. The 180 mg loading dose will be administered as soon as possible by investigation staff after a baseline VerifyNow measurement and after signed informed consent. Patients will be asked to chew, but not to swallow, during at least 40 seconds in presence of investigation staff.
  Drug: ticagrelor (Brilinta) 90 mg tablets, 2 tablets chewed
  Interventions: Drug: Chewed ticagrelor
- Swallowed ticagrelor (Active Comparator): Ticagrelor integral tablet. The 180 mg loading dose will be administered as soon as possible by investigation staff after a baseline VerifyNow measurement is drawn. Patients will swallow the loading dose followed by 25-40 ml of water.
  Drug: ticagrelor (Brilinta) 90 mg tableta, 2 tablets swallowed
  Interventions: Drug: Swallowed ticagrelor

INTERVENTIONS:
Drug: Chewed ticagrelor — Chewed ticagrelor (Brilinta) 90 mg tablets, 2 tablets
  Arms: Chewed ticagrelor
Drug: Swallowed ticagrelor — Swallowed ticagrelor (Brilinta) 90 mg tablets, 2 tablets
  Arms: Swallowed ticagrelor

SUMMARY:
The study aims to determine the pharmacodynamic performance in the first hour measured with verifynow, of the conventional ticagrelor loaded dose versus chewed ticagrelor in patients with acute coronary syndrome treated with percutaneous coronary intervention

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to the emergency department with acute coronary syndrome for percutaneous coronary intervention

Exclusion Criteria:

* Age <18 years
* Known coagulopathy, bleeding diathesis, or active bleeding
* History of recent gastrointestinal or genitourinary bleeding within 2 months
* Previous therapy with clopidogrel, prasugrel, or ticagrelor
* Previous treatment with glycoprotein IIb/IIIa inhibitors or during interventional procedure
* Major surgery within 6 weeks
* History of intracranial bleeding or intracraneal neoplasm
* Suspected aortic dissection
* Chronic obstructive pulmonary disease
* Severe hemodynamic instability or cardiogenic shock
* Resuscitated cardiac arrest
* Use of vitamin K anticoagulants or novel oral anticoagulants (NOACs) within 7 days
* Life expectancy <1 year
* Known severe liver or renal disease, GFR estimated by CKD-EPI <30 ml/min/1.73 m2
* Known HIV treatment
* Hemoglobin <10 g/dL
* Platelet count <100,000/L
* Pregnancy
* Known allergy to ticagrelor
* Refusal to sign informed consent

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity | 1 hour
  Platelet reactivity measured with VerifyNow (PRU)

SECONDARY OUTCOMES:
Efficacy (MACCE) | 30 days
  Composite outcome: made by major adverse cardiac and cerebrovascular events: all-cause death, repeat myocardial revascularization, stroke, myocardial infarction
Composite outcome | 30 days
  Composite outcome: major bleeding, AND nonmajor clinically relevant (NMCR) bleeding both by ISTH definition
Efficacy (long term) | 1 year
  Composite outcome: number of participants with major adverse cardiac and cerebrovascular events (MACCE) (previously defined)
High platelet reactivity on treatment rate | 1 hour
  Inhibition of platelet aggregation (IPA) measured by VerifyNow

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Concepción, Saltillo, Coahuila, Mexico

IPD SHARING:
Plan to Share IPD: No